

## 'ILD in Screening' Research Database

## **Consent Form**

Thank you for reading the information leaflet about the ILD in Screening Study Research Database. If you consent to your information being entered on the database, please read and sign this form **and put your initials in the boxes**.

| 1. | I have read the attached information sheet and have been given a copy to keep. I have been able to ask questions and have had these answered to my satisfaction. |
|---|---|
| 2. | I agree that staff from the ILD in Screening study research team may look at my medical records or contact health professionals responsible for my care to obtain information on my clinical history, investigations and outcome, where relevant to lung disease. |
| 3. | I agree that information about me from the ILD in Screening study can be held on the ILD in Screening study Research Database. |
| 4. | I agree that information from my medical records, including future medical records, about tests or treatment for lung disease can be held on the ILD in Screening Research Database. |
| 5. | I agree that anonymised information from the ILD in Screening Research Database can be released to third parties for use in ethically approved future research. |
| 6. | I understand that my records may be looked at by authorised individuals from the Sponsor for the study and the UK Regulatory Authority in order to check that the study is being carried out correctly. |



| Name of Patient | Date | Signature |
|---|---|---|
| Name of Person Taking Consent | <br>Date | Signature |
| Thank you for agreeing to participate in this study. | | |
| When completed: 1 for patient: | 1 for service file (orig | inal) |